CLINICAL TRIAL: NCT02386982
Title: A Single-centre, Randomized, Open-label, 2-arm, 4-week Treatment Study to Investigate the Beta Cell Function and Related Pharmacodynamics in Type 2 Diabetes Mellitus (T2DM) Patients
Brief Title: Beta Cell Function and Related Pharmacodynamics of HMS5552 in T2DM Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hua Medicine Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMM0103
Record Dates: First submitted 2015-03-05; First posted 2015-03-12 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dorzagliatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HMS5552 dose 1 (Experimental): HMS5552 75mg.Oral administration,twice per day.
  Interventions: Drug: HMS5552
- HMS5552 dose 2 (Experimental): HMS5552 75mg.Oral administration,once per day.
  Interventions: Drug: HMS5552

INTERVENTIONS:
Drug: HMS5552
  Other Names: Sinogliatin

SUMMARY:
This study evaluates the beta cell function, pharmacodynamics, pharmacokinetics, safety and tolerability after 4 weeks treatment of 75mgBID or 75mgQD of HMS5552.

ELIGIBILITY:
Inclusion Criteria:

* Male and female,age 18-65 years
* Has type 2 diabetes mellitus
* BMI 20 to 29kg/m2
* Willingness to adhere to the protocol requirement

Exclusion Criteria:

* Patients with type1 diabetes mellitus
* Received any antidiabetic drug within run-in or during screening
* Hepatic diseases
* Kidney diseases
* Clinical abnormal finding in EVG,labs and physical exams
* Women of child-bearing potential

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
beta cell function | 4 weeks
  will be assessed by change of beta cell function index
HbA1 | 4 weeks
24-hour glucose change | 4 weeks

SECONDARY OUTCOMES:
The study drug concentration in blood samples to be collected after drug administration | 4 weeks
Composite measure of adverse events monitoring, physical examinations,12 lead ECGs, vital sign,and safety laboratory measurement | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The 1st Betuhune Hospital of Jilin University, Changchun, China